CLINICAL TRIAL: NCT02194179
Title: Steady State Bioavailability of 2 Different Nevirapine Extended Release Formulations Compared to Steady State 400 mg of Viramune® (200 mg BID), in HIV-1 Infected Subjects, an Open Label, Non Randomised, Multidose and Multistage Parallel Group Study. (ERVIR)
Brief Title: Bioavailability of 2 Different Nevirapine Extended Release Formulations Compared to Viramune® in HIV-1 Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1489
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

ARMS (9):
- NVP XR 400 mg (KCR 25%) fasted (Experimental)
  Interventions: Drug: NVP XR 400 mg (KCR 25%)
- NVP XR 400 mg (KCR 25%) fed (Experimental)
  Interventions: Drug: NVP XR 400 mg (KCR 25%); Other: high-fat breakfast
- NVP XR 400 mg (KCR 20%) fasted (Experimental)
  Interventions: Drug: NVP XR 400 mg (KCR 20%)
- NVP XR 400 mg (KCR 20%) fed (Experimental)
  Interventions: Drug: NVP XR 400 mg (KCR 20%); Other: high-fat breakfast
- NVP XR 300 mg (KCR 25%) fasted (Experimental)
  Interventions: Drug: NVP XR 300 mg (KCR 25%)
- NVP XR 300 mg (KCR 25%) fed (Experimental)
  Interventions: Drug: NVP XR 300 mg (KCR 25%); Other: high-fat breakfast
- NVP XR 300 mg (KCR 20%) fasted (Experimental)
  Interventions: Drug: NVP XR 300 mg (KCR 20%)
- NVP XR 300 mg (KCR 20%) fed (Experimental)
  Interventions: Drug: NVP XR 300 mg (KCR 20%); Other: high-fat breakfast
- NVP IR 200 mg (Viramune®) (Active Comparator)
  Interventions: Drug: NVP IR 200 mg (Viramune®)

INTERVENTIONS:
Drug: NVP XR 400 mg (KCR 25%)
  Arms: NVP XR 400 mg (KCR 25%) fasted; NVP XR 400 mg (KCR 25%) fed
Drug: NVP XR 400 mg (KCR 20%)
  Arms: NVP XR 400 mg (KCR 20%) fasted; NVP XR 400 mg (KCR 20%) fed
Drug: NVP XR 300 mg (KCR 25%)
  Arms: NVP XR 300 mg (KCR 25%) fasted; NVP XR 300 mg (KCR 25%) fed
Drug: NVP XR 300 mg (KCR 20%)
  Arms: NVP XR 300 mg (KCR 20%) fasted; NVP XR 300 mg (KCR 20%) fed
Other: high-fat breakfast
  Arms: NVP XR 300 mg (KCR 20%) fed; NVP XR 300 mg (KCR 25%) fed; NVP XR 400 mg (KCR 20%) fed; NVP XR 400 mg (KCR 25%) fed
Drug: NVP IR 200 mg (Viramune®)
  Arms: NVP IR 200 mg (Viramune®)

SUMMARY:
The objective was to establish the pharmacokinetic (PK) profile at steady state of two different nevirapine (NVP) extended release (XR) formulations at 300 mg or 400 mg daily (QD) under fasted and fed conditions in comparison with the commercially available NVP immediate release (IR) tablet at 200 mg BID (400 mg/day).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected males or females ≥ 18 and ≤ 60 years of age
* Body mass index 18.5 to 29.9 kg/m2, inclusive
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and local legislation
* Treated with a stable Viramune® BID based regimen since at least 12 weeks prior to study entry. If however, the subject's current Viramune® treatment consists of two 200mg tablets once daily (prescribed off label), the subject is allowed to participate if he/she agrees to switch to Viramune® 200mg twice daily, 14 days before the start of Nevirapine Extended Release.
* An HIV-1 viral load of ≤ 50 c/mL at screening
* Acceptable screening laboratory values that indicate adequate baseline organ function with the following exceptions:

  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)

    ≤2.5 times the upper limit of normal (ULN) (DAIDS Grade 1) or
  * Gamma-glutamyl transferase (GGT) <2.5 times ULN (DAIDS Grade 1)
* Willingness to abstain from alcoholic beverages for 24 hours prior to intensive pharmakokinetic sampling days
* Willingness to abstain from ingesting substances which may alter drug plasma levels by interaction with the cytochrome P450 system during the study
* Willingness to abstain from grapefruit and grapefruit juice, Seville oranges and juice, and St John's wort or milk thistle starting 14 days prior to administration of study medication until the end of the study, and
* Karnofsky performance score ≥70

Exclusion Criteria:

* Current treatment with any PI
* Participation in another trial with an investigational medicine within two months prior to Day 1 of this study
* Serum creatinine levels >1.5 times ULN at screening
* History of acute illness within 60 days prior to Day 1, which would make the subject, in the opinion of the investigator, unsuitable for the trial
* History or evidence of severe illness, malignancy or any other conditions which would make the subjects, in the opinion of the investigator, unsuitable for the trial
* Any evidence of a clinically relevant concomitant disease, including gastrointestinal, hepatic, renal disorders of clinical relevance
* Surgery of the gastrointestinal tract (except appendectomy and herniotomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections other than HIV-1 (e.g. hepatitis B virus (HBV), hepatitis C virus (HCV) co infection: A chronic or acute HBV infections is defined as: HBs Ag positive. Chronic or acute HCV infection is defined as: HCV Ab positive and 1 confirmed positive viral load measurement preceding study entry)
* Alcohol or substance abuse within 6 months prior to screening or during the study
* Inability to comply with protocol requirements
* Screening laboratory values <DAIDS grade 1
* All fertile males or females, and their respective partner(s) not willing to use two forms of effective contraception. A double-barrier method must be used. A double-barrier method is defined as e.g.: 1) a condom with spermicidal jelly or with a foam suppository; 2) a diaphragm with spermicide; or 3) a male condom and a diaphragm
* Female of child-bearing potential who:

  * Has a positive serum pregnancy test at screening,
  * Is breastfeeding,
  * Is planning to become pregnant, or
  * Is not willing to use barrier method protection or require ethinyl estradiol administration
* Any AIDS-defining illness that is unresolved, symptomatic, or not stable on treatment for at least 12 weeks before the screening visit
* HIV-2 infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over the time dosing interval τ) | up to day 22
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over the time dosing interval τ) | up to day 22
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over the time dosing interval τ) | up to day 22

SECONDARY OUTCOMES:
Cmax,ss / Cmin,ss ratio | up to day 22
%PTF (percentage peak-trough fluctuation) | up to day 22
tmax,ss (time from dosing to the maximum concentration of the analyte in plasma at steady state over the time dosing interval τ) | up to day 22
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | up to day 22
Cavg (average measured concentration of the analyte in plasma at steady state) | up to day 22
Number of patients with adverse events (AEs) | up to day 57
Number of patients with clinically relevant changes in clinical laboratory tests | Baseline, up to day 37
Number of patients with abnormal detectable viral load | Baseline, up to day 37
Number of patients with clinically relevant changes in vital signs (blood pressure, pulse rate) | Baseline, up to day 37
Number of patients with clinically relevant changes in 12-lead electrocardiogram (ECG) | Baseline, day 23
Number of patients with clinically relevant changes in physical examination | Baseline, up to day 37
Assessment of tolerability by the investigator on a 4-point scale | up to day 37